CLINICAL TRIAL: NCT05315427
Title: Impact of Music Therapy on Pain in Patients Treated for Advanced Cancer
Acronym: MSPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PROICM 2021-10 OMS; 2021-A02020-41 (Other: ID RCB number of competent autority in France)
Record Dates: First submitted 2022-03-17; First posted 2022-04-07 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Advanced Cancer
Keywords: music therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of the impact of music therapy on the pain of patients (Experimental): One music therapy session
  Interventions: Other: one music therapy session

INTERVENTIONS:
Other: one music therapy session — Edmonton Symptom Assessment System (ESAS) scale (before and after music therapy session), Numerical pain scale (before and after music therapy session)

SUMMARY:
The aim of this study is to assess the impact of music therapy on the pain of patients cared at the Montpellier Cancer Institute (ICM) for advanced cancer in a palliative situation and requiring full hospitalization or on an outpatient basis.

DETAILED DESCRIPTION:
Music therapy is a care practice that falls within the field of support, help and accompaniment therapies. Sound, musical and music are the means used to support, maintain or improve a person's physical and mental health.

The patients involved in the study are patients cared at the ICM for advanced cancer in a palliative situation and requiring full hospitalization or on an outpatient basis.

The aim is to assess the impact of music therapy on the pain of these patients. The patient is proposed to participate in a music therapy session. Before this session, the music therapist will assess the pain and the presence of symptoms with the patient.

Following this exchange, she will define the device best suited to his expectations and his needs and will propose his a relaxation session induced by music.

After the session the music therapist will assess with the patient the pain and the presence of symptoms.

The patient's feelings and satisfaction about this music therapy session as well as his possible wish to participate in another session will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male/female over 18 years old
* Patient cared for at the ICM for advanced cancer followed by the Mobile Palliative and/or Pain Care Team
* Patient with pain score >= 3 (cancer related)
* Patient who accepts a music therapy session
* Patient having expressed his oral non-opposition
* Patient able to communicate
* Patient affiliated to the French Social Security System.

Exclusion Criteria:

* Patient with uncorrected hearing loss to normal
* Patient under guardianship, curatorship or safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Change between before and after music therapy session on patients pain | at day 1 (before and after the music therapy session)
  Evolution of pain assessed by a numerical pain scale ranging from 0 to 10 (10 indicating the highest degree of pain)

SECONDARY OUTCOMES:
Description of symptom management | at day 1 (before and after the music therapy session)
  By the Edmonton Symptom Assessment System scale symptom score. This is a self-assessment scale of the most common symptoms in palliative care:pain, dyspnoea, fatigue, drowsiness, appetite, anxiety, depression, well-being and other possible symptoms. It's a numerical scale ranging from 0 to 10 (with higher scores indicating more severe symptoms).
  The Edmonton Symptom Assessment System scale allows to:
  * Detect the symptoms present, quantify them and follow their evolution
  * Validate with the patient the symptoms that bother him and that he wishes to be treated as a priority
  * Communicate quickly between the different professionals involved in the treatment.
Patient wishing a second session of music therapy | at day 1 (after the music therapy session)
  Proportion of Patient wishing a second session of music therapy
Patient satisfaction of the music therapy session | at day 1 (after the music therapy session)
  Assessment of the satisfaction of the music therapy session. Assessment made by a numerical scale ranging from 0 to 10 (10 indicating high satisfaction)
Agreement to participate in the study | at inclusion
  Proportion of patients agreeing to participate among the eligible patients to whom the study was proposed

CONTACTS AND LOCATIONS:
Overall Officials: Caroline GALLAY, Study Chair — Institut du Cancer de Montpellier - Val d'Aurelle
Locations (1):
- Institut du Cancer de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siedliecki SL, Good M. Effect of music on power, pain, depression and disability. J Adv Nurs. 2006 Jun;54(5):553-62. doi: 10.1111/j.1365-2648.2006.03860.x. PMID 16722953
- [Background] Beck SL. The therapeutic use of music for cancer-related pain. Oncol Nurs Forum. 1991 Nov-Dec;18(8):1327-37. PMID 1762973
- [Background] Huang ST, Good M, Zauszniewski JA. The effectiveness of music in relieving pain in cancer patients: a randomized controlled trial. Int J Nurs Stud. 2010 Nov;47(11):1354-62. doi: 10.1016/j.ijnurstu.2010.03.008. Epub 2010 Apr 18. PMID 20403600
- [Background] Krishnaswamy P, Nair S. Effect of Music Therapy on Pain and Anxiety Levels of Cancer Patients: A Pilot Study. Indian J Palliat Care. 2016 Jul-Sep;22(3):307-11. doi: 10.4103/0973-1075.185042. PMID 27559260
- [Background] Alcantara-Silva TR, de Freitas-Junior R, Freitas NMA, de Paula Junior W, da Silva DJ, Machado GDP, Ribeiro MKA, Carneiro JP, Soares LR. Music Therapy Reduces Radiotherapy-Induced Fatigue in Patients With Breast or Gynecological Cancer: A Randomized Trial. Integr Cancer Ther. 2018 Sep;17(3):628-635. doi: 10.1177/1534735418757349. Epub 2018 Apr 10. PMID 29633652
- [Background] Boyde C, Linden U, Boehm K, Ostermann T. The Use of Music Therapy During the Treatment of Cancer Patients: A Collection of Evidence. Glob Adv Health Med. 2012 Nov;1(5):24-9. doi: 10.7453/gahmj.2012.1.5.009. Epub 2012 Nov 1. PMID 27257528
- [Background] Bradt J, Dileo C, Magill L, Teague A. Music interventions for improving psychological and physical outcomes in cancer patients. Cochrane Database Syst Rev. 2016 Aug 15;(8):CD006911. doi: 10.1002/14651858.CD006911.pub3. PMID 27524661
- [Background] Lesiuk T. The Development of a Mindfulness-Based Music Therapy (MBMT) Program for Women Receiving Adjuvant Chemotherapy for Breast Cancer. Healthcare (Basel). 2016 Aug 9;4(3):53. doi: 10.3390/healthcare4030053. PMID 27517966